CLINICAL TRIAL: NCT03271957
Title: Relation of Ultrasound Parameters Associated to Labor Progression and Manual Rotation's Success in Persistent Occiput Posterior Position
Brief Title: Manual Rotation in Persistent Occiput Posterior Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ana Catarina Reis de Carvalho (Other)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor-Investigator, Ana Catarina Reis de Carvalho, Resident, University of Lisbon
Organization: University of Lisbon (Other)
Other Study IDs: ManualRotationULisbon
Record Dates: First submitted 2017-07-17; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Manual Rotation of A Liveborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Manual rotation — Rotation of the fetal head to an anterior position at time of fuel dilation that is part of routine care

SUMMARY:
Is part of routine obstetric care to attempt a manual rotation in all fetus that are in a persistent OP at delivery. Nevertheless, little is known about the success of this intervention or about the relation of some ultrasound measures with the outcome.

DETAILED DESCRIPTION:
Persistent OP at delivery occurs in approximately 10% of fetuses and studies have shown an increase in short-term and long-term maternal and fetal complications such as prolonged labour, maternal exhaustion, fetal distress, instrumental delivery, caesarean delivery and severe perineal tears. Manual rotation of the fetal occiput to OA position has been described as a safe and effective intervention in the setting of labour arrest but evidence is limited. Therefore, the investigators aim to evaluate:

1. The success of manual rotation of the fetal occiput in OP in 2nd stage of labour; The relation of progression angle (PA) accessed by ultrasound and the success of manual rotation; This is as prospective study with a sample size calculated of 50 participants.

1. º Identify an OP position during digital examination in the first evaluation at full cervical dilatation (t=0)
2. º Get informed consent from the pregnant woman.
3. º Wait for the first urge to push or T=30 m (multiparous) or T=60 (nulliparous)
4. º Confirm fetal head position by ultrasound and measure PA.
5. º Attempt a manual rotation to anterior position accordingly to the protocol.
6. º Confirm fetal head position by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* >37 weeks of pregnancy
* Fetus in cephalic presentation
* Fetal weight estimation P10-90
* Fetal head in a posterior position in the moment of full cervical dilatation.

Exclusion Criteria:

- do not give or do not be able to give written consent

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: All pregnant women in the delivery room that fulfill the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-02-27 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Success of manual rotation of the fetal occiput in OP in 2nd stage of labour | This outcome will be measure immediately after the attempt of manual rotation
  After the attempt of manual rotation we will confirm if the fetal occiput, initially in Occiput-posterior (OP) position, is now in Occiput-anterior position (successful rotation) or if is still in OP position (unsuccessful rotation). This confirmation will be made through ultrasound observation.

SECONDARY OUTCOMES:
Impact of ultrasound measures (progression angle (PA) and dorsal fetal position) | The PA and dorsal fetal position will be measure after the diagnose of full dilatation when occurs the first urge to push or 30 minutes after the diagnose of full dilatation (multiparous) or 60 minutes after the diagnose of full dilatation (nulliparous)
  The relation of PA and dorsal fetal position accessed by ultrasound and the success of manual rotation;

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Clode, MD, Study Director — Obstetrics' Director
Locations (1):
- Departamento de Obstetrícia, Ginecologia e Medicina da Reprodução, Centro hospitalar lisboa norte, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No